CLINICAL TRIAL: NCT04578275
Title: STRATIFY TRIAL: Atrial Fibrillation Stratification Based on the Arrhythmia Perpetuation Mechanisms.
Brief Title: Atrial Fibrillation Stratification Based on the Arrhythmia Perpetuation Mechanisms
Status: Completed | Type: Observational
Sponsor: Felipe Atienza (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Sponsor-Investigator, Felipe Atienza, Head of cardiovascualar research and training, Cardiology Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: STRATIFY-AF
Record Dates: First submitted 2020-03-05; First posted 2020-10-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diagnostic strategy using ECGI — Procedure: Drug treatment, CVE, Pulmonary vein ablation isolation according to treatment guidelines and investigators discretion.
  ECGI: customized body surface mapping (57 electrodes) at the inclusion in the study, after treatment assignment and prior to AF ablation procedure.

SUMMARY:
Atrial fibrillation treatments have a limited efficacy and often cause long-term side effects. This study aims to develop and validate an ECGI system to risk stratification in patients with persistent AF, identifying the mechanisms responsible for the maintenance and the best treatment for ending it.

DETAILED DESCRIPTION:
The MAIN GOAL of this project is to clinically validate the technology for the noninvasive identification of the mechanisms responsible for maintenance of AF using ECGI. To achieve this goal, the investigators will analyze the efficacy of different treatment options in persistent AF patients as a function of the results of the ECGI. Mainly, patients will be evaluated attending to the complexity of the patterns obtained. Moreover, the investigators will evaluate the treatment benefit of performing guided-ablation in conjunction with pulmonary vein isolation as compared to pulmonary vein isolation only. These analyses will be performed in patients with persistent AF arriving at the clinic to determine treatment options. AF outcomes following the treatment assigned therapy will be evaluated at 6 months and 1 year after.

These parameters are obtained from the ECGI map: histogram of rotors (number of rotors and location), Highest and Lowest Dominant Frequency (Hz), rotor duration (ms), simultaneous rotors (number of rotors) and signal entropy (normalized).

Wide antrum circumferential pulmonary vein isolation with demonstration of bidirectional block will be performed using standard cooled-tip radiofrequency catheters or cryoballoon catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF symptomatic and refractory to at least one antiarrhythmic medication arriving in atrial fibrillation to the AF clinic.
* Patients with paroxysmal AF undergoing AF ablation in whom AF was induced at the EP laboratory.
* Patients with persistent AF or long-term persistent AF attending the AF clinic.
* Patients must be able and willing to provide written informed consent to participate in the study.
* Prior anticoagulation for> 4 weeks or transesophageal echocardiogram excluding intracardiac thrombi.

Exclusion Criteria:

Inclusion Criteria:

* Patients with paroxysmal AF symptomatic and refractory to at least one antiarrhythmic medication arriving in atrial fibrillation to the AF clinic.
* Patients with paroxysmal AF undergoing AF ablation in whom AF was induced at the EP laboratory.
* Patients with persistent AF or long-term persistent AF attending the AF clinic.
* Patients must be able and willing to provide written informed consent to participate in the study.
* Prior anticoagulation for> 4 weeks or transesophageal echocardiogram excluding intracardiac thrombi.

Exclusion Criteria:

* Patients with inadequate anticoagulation levels, left atrial thrombus, tumor, or another abnormality which precludes catheter introduction on TEE prior to the procedure.
* Patients with moderate-to-severe mitral regurgitation.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin.
* Patients who are or may potentially be pregnant.
* Current enrollment in another investigational drug or device study.
* Pacemaker or Implantable Cardioverter Defibrillator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients manifesting atrial fibrillation at the AF clinic
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
ECGI calculation of frecuency maps(Hz) | 12 months post-first intervention
  Freedom from atrial fibrillation treated according to the ESC/AHA Atrial Fibrillation Guidelines in relation to the ECGI AF complexity score
ECGI calculation of frecuency of rotor maps | 12 months post-first intervention
  number of rotors mesasured Atrial Fibrillation Guidelines in relation to the ECGI AF complexity score
ECGI AF complexity score calculated from the results of 1 and 2 to evaluate AF freedom from atrial fibrilation | 12 months post-first intervention
  score calculated from the results of 1 and 2 to evaluate AF freedom from atrial fibrilation Atrial Fibrillation Guidelines in relation to the ECGI AF complexity score

SECONDARY OUTCOMES:
Freedom from atrial fibrillation treated according to the ESC/AHA atrial fibrillation Guidelines evaluated in binary(0:AF Freedom;1:AF) | 12 months post-first intervention
Freedom from atrial fibrillation in patients undergoing rhythm control drug treatment. | at 6 and 12 months
Freedom from atrial fibrillation and other atrial arrhythmias in patients undergoing surgical AF ablation. | at 6 and 12 months
ECGI calculations of Highest Dominant Frecuency(Hz) | during ablation procedure and 12 months after
ECGI calculations of Lowest Dominant Frecuency(Hz) | during ablation procedure and 12 months after
ECGI calculations of Rotor duration from rotor maps(ms) | during ablation procedure and 12 months after
ECGI calculations of simultaneus number of rotors from rotor maps(ms) | during ablation procedure and 12 months after
Ablation procedure duration | Duration of ablation procedure
Electrophysiological characteristics of the Atrial fibrillation complexity | Inclusion, rhythm vs rate treatment, ablation
  Atrial fibrillation characteristics will be assesed according to the parameters obtained from ECGi calculations. These parameters are obtained from the frecuency maps(Hz) and histogram of rotors(number of rotors and location) and include : Highest and Lowest Dominant Frecuency(Hz), rotor duration(ms) and simultaneous rotors(number of rotors)
Electroanatomic reconstruction and recordings of electrical activity | During ablation procedure
  a three-dimensional reconstruction of atrium and coronary sinus is obtained using high density catheters and an electroanatomic navigation system.
Fluoroscopy time | During ablation procedure, in minutes
Trained Neural Network based on ECGI signals | 6 and 12 month post-ablation outcome prediction

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No